CLINICAL TRIAL: NCT03697122
Title: Heated Humidified Breathing Circuit Rewarming in Hypothermic Post Cardiopulmonary Bypass Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100711
Record Dates: First submitted 2018-09-27; First posted 2018-10-05 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Hypothermia; Rewarming
Keywords: Cardiopulmonary bypass; Afterdrop; Deep Hypothermic Circulatory Arrest; Heated Humidified Breathing Circuit
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: The intervention group has only one arm. All patients will use active warming via traditional methods (ie forced air warming blankets) and Heated Humidified breathing circuits (HHBC) via ANAPOD Heated Humidification System® (ANAPOD). Those patients will be matched with a retrospective historical cohort of patients that received active warming via traditional methods only (forced air warming blankets).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- HHBC and Forced Air Warming (Experimental): Patients admitted to intensive care unit hypothermic (≤ 35 C) following surgical procedures involving cardiopulmonary bypass. Will be rewarmed with heated humidified breathing circuits (ANAPOD) and standard forced air warming blankets.
  Interventions: Device: Heated Humidified Breathing Circuit and Forced Air Blanket

INTERVENTIONS:
Device: Heated Humidified Breathing Circuit and Forced Air Blanket — Heated humidified breathing circuits (ANAPOD) will be set up and managed by respiratory therapist in standard fashion defined by the manufacturer. Temperate will be set at 41C.
  Forced air warming blankets will be set at 42C for duration of rewarming.
  Other Names: ANAPOD

SUMMARY:
Hypothermia on admission to the intensive care unit (ICU) following cardiopulmonary bypass (CPB) is common. The investigators propose that rewarming hypothermic (≤ 35 C) patients admitted to the intensive care unit following procedures using CPB with heated humidified breathing circuits (HHBC) in addition to conventional forced air warming blankets will shorten time to normothermia. Secondarily it may shorten time to extubation, improve coagulopathy, and metabolic derangements seen with hypothermia.

DETAILED DESCRIPTION:
Hypothermia on admission to the intensive care unit (ICU) following cardiopulmonary bypass (CPB) is common. Cooling and rewarming during CPB and deep hypothermic circulatory arrest (DHCA) takes considerable time and contributes to the post-procedural coagulopathy and physiologic perturbations. Core body parts (trunk and head) rewarm more quickly than peripheral parts (extremities). After disconnecting from CPB the body is allowed to self equilibrate. The normal vasoconstriction response is impaired by the administered anaesthesia. Hence, heat distribution takes place from the warm core to the colder periphery. This causes an afterdrop: a decrease in the temperature of the core organs. After-drop may contribute to post-operative complications such as shivering, coagulopathy, increased myocardial stress, increased wound infections, metabolic acidosis, delayed extubation and prolonged ICU length of stay (LOS).

The use of the active warming via traditional methods (ie forced air warming blankets) and Heated Humidified breathing circuits (HHBC) via ANAPOD Heated Humidification System® (ANAPOD) may shorten time to normothermia. Secondarily it may shorten time to extubation, improve coagulopathy, and metabolic derangements seen with hypothermia.

Sample and Study Design- The investigators will prospectively collect data for 14 enrolled non-patients who will receive active warming via both forced air warming blankets and Heated Humidified breathing circuits (HHBC). Retrospective data will be obtained retrospectively for 28 matched patients from two years prior to initiation of the trial, who received warming only via forced air warming blankets.

Data Collection Plan- Data will be extracted and collected by the Duke Department of Anesthesiology IT analyst, who will review and extract information from the patient's chart via Epic/ Maestro Care, or manually if necessary.

Data Evaluation- Descriptive statistics will be used to evaluate patient demographics and clinical characteristics. Descriptive statistics will be summarized as mean ± (SD) or median (interquartile range) for continuous variables and group frequencies (%) for dichotomous or categorical variables.

As all patients are expected to achieve normothermia within the study period, the primary outcome of time to normothermia will be analyzed as a numeric outcome variable. Following validation of distributional assumptions the investigators will compare the time to normothermia between the two groups via t-test or Wilcoxon rank sum test as appropriate. It is expected that the patients will reach normothermia between 45 minutes and 6 hours after admission to the ICU.

By using a 2:1 matching ratio and a moderate level of variability (SD=1.3 hours) a study of 14 prospectively enrolled patients and 28 retrospectively matched patients would attain 82% power to detect a 1.25 hour difference between time to normothermia in the prospective group (active warming via traditional methods (ie forced air warming blankets) and Heated Humidified breathing circuits (HHBC) via ANAPOD Heated Humidification System® (ANAPOD), and the retrospective group (active warming via traditional methods (ie forced air warming blankets only) at alpha level 0.05.

Secondary numeric outcomes such as time to extubation, time to normal PH, and coagulopathy lab values will be analyzed by t-test or Wilcoxon rank sum test as appropriate. Differences in categorical outcomes between treatment groups will be analyzed via chi-square or fisher exact tests. As the patients will be matched on key confounders no further adjustment is expected to be necessary, so the moderate sample size should not limit the primary analysis. Potential subgroup analysis may be conducted in an exploratory analysis to determine if the treatment effect of ANAPOD warming is different by procedure type or patient/surgical characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Admission to intensive care unit following surgical procedure involving cardiopulmonary bypass.
* Admission temperature ≤ 35.0 C.

Exclusion Criteria:

* Patients placed on extracorporeal membrane oxygenation intra-operatively, or during first 24 hours after ICU admission.
* Any additional surgical procedures in the first 24 hours days after initial surgery e.g. Chest exploration for bleeding, Open Chest, Non-cardiac surgery such as colectomy for ischemic gut, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Negmeldeen Mamoun, MD, Principal Investigator — Duke Univeristy Hospital Anesthesia Department
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- HHBC and Forced Air Warming: Patients admitted to intensive care unit hypothermic (≤ 35 C) following surgical procedures involving cardiopulmonary bypass. Will be rewarmed with heated humidified breathing circuits (ANAPOD) and standard forced air warming blankets.
  Heated Humidified Breathing Circuit and Forced Air Blanket: Heated humidified breathing circuits (ANAPOD) will be set up and managed by respiratory therapist in standard fashion defined by the manufacturer. Temperate will be set at 41C.
  Forced air warming blankets will be set at 42C for duration of rewarming.
Period: Overall Study
Arm/Group | HHBC and Forced Air Warming
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Temperature at ICU admission [Median (Inter-Quartile Range); unit: Degrees Celsius] | 34 [34 to 35]

OUTCOME MEASURES:

1. Primary Outcome: Time to Normothermia
Description: Core temperature normothermia defined as >=36.5 C.
Time Frame: up to 24 hours post admission to intensive care unit
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
hours | 4.4 [3.5 to 5.5]

2. Secondary Outcome: Time to Extubation
Description: Time from admission to time of extubation. Followup was truncated at 24 hours and if patient had not been extubated at that time they were assigned a value of 24 hours.
Time Frame: up to 24 hours post admission to intensive care unit
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
hours | 5.4 [4.9 to 8.0]

3. Secondary Outcome: Coagulopathy as Measured by Need for Transfusion of Blood Product
Description: Assessed via number of transfusions of red blood cells, fresh frozen plasma, platelets, cryoprecipitate.
Time Frame: 24 hours post admission to intensive care unit
Measure: Median (Full Range); unit: Units transfused
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
Units transfused | 0 [0 to 5]

4. Secondary Outcome: Metabolic Derangement as Measured by Time to Normal pH
Description: Assessed via blood gas analysis. Normal pH defined as 7.35-7.45.
Time Frame: up to 24 hours post admission to intensive care unit
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
hours | 0.4 [0.2 to 4.8]

5. Secondary Outcome: Number of Subjects With Abnormal Coagulopathy as Measured by Laboratory Assessment of Prothrombin Time
Description: Laboratory assessment of Prothrombin Time with normal defined as 9.5-13.1 seconds.
Time Frame: 24 hours post admission to intensive care unit
Measure: Count of Participants; unit: Participants
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
Participants | 12

6. Secondary Outcome: Number of Subjects With Abnormal Coagulopathy as Measured by Laboratory Assessment of INR
Description: Laboratory assessment of international normalised ratio (INR) with normal defined as 0.9-1.1.
Time Frame: 24 hours post admission to intensive care unit
Measure: Count of Participants; unit: Participants
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
Participants | 12

7. Secondary Outcome: Number of Subjects With Abnormal Coagulopathy as Measured by Laboratory Assessment of Act Partial Thromboplastin Time
Description: Laboratory assessment of Act Partial Thromboplastin Time with normal defined as 26.8-37.1 seconds.
Time Frame: 24 hours post admission to intensive care unit
Measure: Count of Participants; unit: Participants
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
Participants | 10

8. Secondary Outcome: Number of Subjects With Abnormal Coagulopathy as Measured by Laboratory Assessment of Fibrinogen.
Description: Laboratory assessment of fibrinogen levels with normal defined as 213-435 mg/dL.
Time Frame: 24 hours post admission to intensive care unit
Measure: Count of Participants; unit: Participants
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
Participants | 5

9. Secondary Outcome: Number of Subjects With Abnormal Coagulopathy as Measured by Laboratory Assessment of Platelet Count
Description: Laboratory assessment of platelet count with normal defined as 150 - 450 x10ˆ9/L.
Time Frame: 24 hours post admission to intensive care unit
Measure: Count of Participants; unit: Participants
Arm/Group | HHBC and Forced Air Warming
Number analyzed (Participants) | 14
Participants | 7

ADVERSE EVENTS:
Time Frame: From ICU admission to hospital discharge (ranged between 5 and 9 days)
Arm/Group | HHBC and Forced Air Warming
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HHBC and Forced Air Warming (N=14)
Complete Heart Block (Cardiac disorders) | 1 (1)
Hemorrhagic Stroke (Vascular disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HHBC and Forced Air Warming (N=14)
Atrial Fibrillation (Cardiac disorders) | 5 (5)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Complete Heart Block (Cardiac disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT03697122/Prot_SAP_000.pdf